CLINICAL TRIAL: NCT07345403
Title: GENECARD - the Use of Genetic, Epigenetic, Metabolomic, Proteomic and Microbiotic Markers, Image and Voice Biomarker Analyses, and Pre- and Intraoperative Clinical Data - to Predict Early Complications After Cardiac Surgery.
Acronym: GENECARD
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Collaborators: Politechnika Gdańska (Unknown); University of Gdańsk (Unknown); Pomeranian Medical University Szczecin (Other); Silesian University of Medicine (Other); AGH University of Science and Technology, Krakow, Poland (Unknown)
Responsible Party: Principal Investigator, Maciej M. Kowalik, MD, PhD, DSc, Principal Investigator, Medical University of Gdansk
Other Study IDs: KB/470/2025; 064/2025 (Other: University Clinical Center (Uniwersyteckie Centrum Kliniczne; UCK) Gdańsk, Poland)
Record Dates: First submitted 2025-12-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Delirium (POD); Postoperative Bleeding; Acute Kidney Injury; Atrial Fibrillation (AF); Vasoplegia
Keywords: Cardiac Surgery; Postoperative Complications; Atrial Fibrillation; Acute Kidney Injury; Postoperative Delirium; Vasoplegia; Biomarkers; Multi-omics; Risk Prediction; Epigenetics; genetics; microbiota; metabolomics
MeSH Terms: conditions — Emergence Delirium; Postoperative Hemorrhage; Acute Kidney Injury; Atrial Fibrillation; Vasoplegia; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples With DNA — The study will retain the following biospecimens collected before and after cardiac surgery:
  Peripheral blood samples, including whole blood, plasma/serum, and PBMCs for:
  Genetic analysis (targeted SNP panels; potential NGS/WGS), Epigenetic profiling (DNA methylation), Transcriptomics (RNA-seq), Proteomic and metabolomic testing, Routine laboratory biomarkers (e.g., creatinine, NGAL, cystatin C, KIM).
  Urine samples for short-chain RNA (scRNA) transcriptomic analyses and metabolomic profiling (pre- and postoperative).
  Stool samples for microbiota and microbiome studies, including bacterial fractions, extracellular vesicles, and metabolite fractions, analyzed with GC-MS and LC-MS/MS and via metagenomic sequencing.
  Digital biospecimens: non-invasive voice and video recordings collected to identify acoustic and image biomarkers of postoperative delirium.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elective Cardiac Surgery Patients: Adult men and women (≥18 years) undergoing elective cardiac surgery who provide informed consent are enrolled. Patients with a history of, or planned, solid organ or bone marrow transplantation are excluded. All participants are followed prospectively during and after surgery to determine the occurrence of early postoperative complications, including new-onset atrial fibrillation, acute kidney injury, postoperative delirium, vasoplegia, and postoperative bleeding, as well as in-hospital and 30-day mortality, duration of mechanical ventilation, and ICU and hospital length of stay.
  Interventions: Other: Multi-Omics Data and Clinical Data Collection

INTERVENTIONS:
Other: Multi-Omics Data and Clinical Data Collection — Collection of blood, urine, stool, imaging data, intraoperative data, and non-invasive digital recordings (voice and video) for genetic, epigenetic, transcriptomic, proteomic, metabolomic, microbiome, laboratory, and clinical analyses. No therapeutic intervention is given. All procedures involve observational data and biospecimen collection before, during, and after elective cardiac surgery.
  Other Names: Biological Sample Collection

SUMMARY:
The goal of this observational cohort study is to prove whether genetic, epigenetic, transcriptomic, proteomic, metabolomic, imaging, voice, and clinical markers can improve prediction of early complications after cardiac surgery in adult patients.

The main questions it aims to answer are:

Which biological and clinical markers are associated with: new-onset atrial fibrillation (NOAF), acute kidney injury (AKI), postoperative delirium (POD), vasoplegia, postoperative bleeding and 30-day mortality? Can combining these markers improve early prediction of postoperative complications compared with current clinical risk scores?

Researchers will analyze a wide range of data collected before, during, and after cardiac surgery and compare patients who develop early complications with those who do not to identify risk factors and early biomarkers.

Participants will:

Provide biological samples (blood, urine, stool) before and after surgery for genetic, epigenetic, transcriptomic, proteomic, metabolomic, microbiome, and laboratory testing.

Undergo standard preoperative and intraoperative imaging and clinical assessments.

Allow collection of clinical data related to postoperative outcomes (For some participants) have voice and video recordings performed to help identify early signs of postoperative delirium.

This study aims to improve early detection of postoperative complications and support development of personalized diagnostic and treatment strategies for patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Single-center, prospective, translational, observational cohort study designed to identify markers that predict early postoperative complications in adult patients undergoing elective cardiac surgery. The study will analyze genetic, epigenetic, transcriptomic, proteomic, metabolomic, microbiome, imaging, voice, and detailed clinical data collected before, during, and after surgery. Approximately 2,000-3,000 participants will be enrolled between 2026 and 2029.

Study Objectives

The main objective is to determine whether selected biological and clinical markers can predict early postoperative complications, including:

New-onset atrial fibrillation (NOAF), Acute kidney injury (AKI), Postoperative delirium (POD), Vasoplegia, Postoperative bleeding 30-day mortality.

The study will use current clinical definitions: NOAF per ESC guidelines, AKI per KDIGO criteria, and POD per DSM-V, as well as validated delirium scales such as CAM-ICU or DOSS. Postoperative bleeding will be defined as >1000 mL drainage in 24 hours or the need for surgical re-exploration.

Secondary outcomes include in-hospital mortality, 30-day mortality, duration of mechanical ventilation, ICU length of stay, and total postoperative hospital length of stay.

Participants

Eligible participants are adult men and women undergoing elective cardiac surgery who provide informed consent. Exclusion criteria are age <18 years, lack of consent, and prior or planned organ or bone marrow transplantation.

Data and Sample Collection

The study will collect a broad set of data and biological materials, including:

Clinical data: detailed medical history, epidemiologic factors, disease history, physical exam parameters, perioperative clinical data, and postoperative complication data.

Genetic analysis: targeted sequencing of selected SNPs associated with primary outcomes using PCR-based arrays or NGS/WGS. DNA from PBMCs will be collected from all participants, with potential additional sequencing pending external funding. A replication cohort of 525 patients from the INFLACOR study will be used for confirmatory analyses.

Epigenetic profiling: genome-wide epigenetic marker profiling from PBMCs in matched case-control subgroups (approximately n=300 per group) for participants who develop primary outcomes. DNA methylation will be analyzed to develop an epigenetic risk index and integrated with genetic and clinical data.

Transcriptomics: RNA-seq of PBMCs collected before surgery, as well as short-chain RNA (scRNA) profiling from urine samples collected pre- and postoperatively to identify early markers of AKI.

Proteomics and metabolomics: untargeted and targeted analyses of plasma collected preoperatively and at two postoperative time points (6 hours and postoperative day 3). These analyses aim to identify and validate early biomarkers of primary complications.

Laboratory diagnostics: serial measurement of selected laboratory markers relevant to early complications, such as serum creatinine, NGAL, cystatin C, and novel biomarkers (e.g., KIM) using ELISA.

Microbiota and microbiome: metabolomic and metagenomic sequencing analyses on fractionated stool samples to characterize gut bacterial composition, extracellular vesicles, and metabolite profiles, using GC-MS and LC-MS/MS.

Imaging data: routine preoperative imaging including transthoracic echocardiography (TTE) and coronary angiography.

Voice and video biomarkers: for participants developing POD, continuous bedside-acquired video, audio, and sensor data will be analyzed to identify voice and image biomarkers (e.g., MFCC parameters) associated with prodromal delirium. Machine-learning models will be developed to support real-time detection of POD-related features.

Analytical Approach

The study will use multistage regression, machine-learning techniques, and AI-based modeling to identify predictors of both primary and secondary outcomes. Analyses will integrate genetic, environmental, preoperative, and intraoperative factors. One aim is to enhance existing clinical risk calculators for postoperative morbidity and mortality, such as STS-ACSD and EuroSCORE. The study expects improved discrimination of predictive models, targeting ROC-AUC values >0.9 for mortality and >0.8 for morbidity.

A polygenic risk score will also be developed to evaluate genetic contribution to variation in primary outcomes.

Expected Impact

The integrated multi-omics and clinical approach is expected to identify new pathophysiological mechanisms underlying early postoperative complications and potentially support development of novel preventive therapies. The study aims to facilitate personalized perioperative diagnostic and therapeutic strategies by improving early identification of high-risk patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Undergoing elective cardiac surgery
* Able and willing to provide informed consent

Exclusion Criteria:

* Age below 18 years
* Lack of informed consent
* Prior or planned solid organ transplantation
* Prior or planned bone marrow transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective cardiac surgery at a single center. Participants include men and women who consent to provide clinical data and biospecimens for analysis. Individuals under 18 years of age or with prior or planned organ or bone marrow transplantation are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
New-onset atrial fibrillation (NOAF) | From end of surgery until hospital discharge, up to 14 days.
  Occurrence of new-onset atrial fibrillation after cardiac surgery, defined according to current ESC guidelines, using clinical data, ECG and centrally recorded rhythm data.
Acute kidney injury (AKI) | From end of surgery until hospital discharge, up to 14 days.
  Occurrence of acute kidney injury after cardiac surgery, defined according to KDIGO criteria, using serial laboratory measurements (including serum creatinine and other kidney biomarkers).Early postoperative period after cardiac surgery during index hospitalization.
Postoperative delirium (POD) | From end of surgery until hospital discharge, up to 14 days.
  Occurrence of postoperative delirium after cardiac surgery, defined according to DSM-V criteria and assessed with validated delirium scales (e.g., CAM-ICU or DOSS), clinical observation, and supporting data (including voice and image recordings in selected patients).
Vasoplegia | Perioperative period and postoperative hospitalization, up to 14 days.
  Occurrence of vasoplegia after cardiac surgery, identified from perioperative and postoperative hemodynamic and clinical data according to prespecified criteria in the protocol.
Postoperative bleeding | Within 24 hours after surgery and during hospitalization for re-exploration, up to 14 days.
  Occurrence of significant postoperative bleeding after cardiac surgery, defined as blood loss >1000 mL in chest drains within 24 hours or the need for surgical re-exploration due to bleeding.

SECONDARY OUTCOMES:
In-hospital mortality | From date of surgery until hospital discharge or death, up to 14 days.
  Death from any cause occurring during the index hospitalization after cardiac surgery.
30-day mortality | 30 days after surgery.
  Death from any cause within 30 days after cardiac surgery, assessed through hospital records and follow-up.
Duration of mechanical ventilation | From end of surgery until final extubation, up to 7 days.
  Total duration of postoperative invasive mechanical ventilation, measured in hours, based on clinical and ICU records.
ICU length of stay | From ICU admission after surgery until ICU discharge, up to 7 days.
  Duration of postoperative stay in the intensive care unit, measured in days, based on clinical records.
Postoperative hospital length of stay | From date of surgery until hospital discharge, up to 14 days.
  Total length of postoperative hospitalization, measured in days, based on clinical records.

CONTACTS AND LOCATIONS:
Overall Officials: Maciej M Kowalik, MD, PhD, Dsc, Study Director — Medical University of Gdansk, Department of Anesthesiology and Intensive Care; Radosław Owczuk, Prof. dr hab., Study Chair — Medical University fo Gdańsk, Department of Anetshesiology and Intensive Care; Kowalik M Kowalik, MD, PhD, Dsc, Principal Investigator — Medical University of Gdansk, Department of Anesthesiology and Intensive Care
Locations (1):
- University Clinical Centre Gdansk, Department of Anaesthesiology and Intensive Care, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual data planed for sharing will include:
  1. anamnesis and structured forms derived data
  2. comorbdities and chronic therapies
  3. laboratory results of blood, urine and other bio specimen exams
  4. genotyped SNP's associated with primary outcome measures
  5. others
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 6 months after starting the recruitment and ending 3 years after last participant recruited.
Access Criteria: Data are planned to be set for open access without restrictions.
URL: https://zenodo.org/